CLINICAL TRIAL: NCT05884658
Title: vNOTEsHC: Hysterectomy by Transvaginal Natural Orifice Transluminal Endoscopic Surgery Versus or Laparoscopic Hysterectomy: a Randomized Controlled Trial
Brief Title: Hysterectomy by Transvaginal Natural Orifice Transluminal Endoscopic Surgery Versus or Laparoscopic Hysterectomy
Acronym: vNOTESHC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21PH265; 2023-A01013-42 (Other: ANSM)
Record Dates: First submitted 2023-05-04; First posted 2023-06-01 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Hysterectomy, Vaginal
Keywords: natural orifice transluminal endoscopy system; large uteri
MeSH Terms: interventions — Hysterectomy

STUDY DESIGN:
Intervention Model Description: prospective, multicenter, randomized, parallel-group, non-inferiority open superiority study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic hysterectomy (Active Comparator): Laparoscopic Hysterectomy will be performed in a standardized manner with or without surgical robot
  Interventions: Procedure: laparoscopic hysterectomy
- natural vaginal orifice transluminal endoscopic system for hysterectomies (vNOTES) (Experimental): Vaginal hysterectomy will be performed in a standardized manner using transluminal endoscopic system
  Interventions: Procedure: vNOTES : natural vaginal orifice transluminal endoscopic system for hysterectomies

INTERVENTIONS:
Procedure: vNOTES : natural vaginal orifice transluminal endoscopic system for hysterectomies — hysterectomy via the vaginal approach by vNOTES (natural vaginal orifice transluminal endoscopic system for hysterectomies)
  Arms: natural vaginal orifice transluminal endoscopic system for hysterectomies (vNOTES)
Procedure: laparoscopic hysterectomy — laparoscopic hysterectomy uses a standardized procedure with or without surgical robot
  Arms: laparoscopic hysterectomy

SUMMARY:
In France, there are approximately 62,000 hysterectomies per year, 70% of which are benign. It is the most frequent surgical procedure in gynecology.

Hysterectomies are performed via 3 routes: laparotomy, laparoscopy or vaginal route.

This choice of approach is particularly important in the case of large uteri (50% of uteri > 280g), which increase the risks of laparoconversion and bladder injury (NP3).

The vaginal route reduces the operating time and postoperative pain. Laparoscopy allows a better anatomical view and easier access to the neighbouring organs, which makes it the preferred approach, especially for young surgeons and when the uterus is large. However, the laparoscopic route is associated with an increase in the rate of conversion to laparotomy according to the volume of the uterus, as well as the rate of general per and postoperative complications compared with vaginal hysterectomy for uteri > 280 g. In a meta-analysis comparing laparoscopy and vaginal hysterectomy, the total prevalence of perioperative complications according to the classification of Clavien and Dindo was 27%. For large uteruses, complications by the vaginal route amounted to 15% and those by the laparoscopic route to 37.5%.

The data are not sufficient to give preference to one or other of the approaches, but for benign pathologies, for large uteri (>280 g), the minimally invasive laparoscopic or vaginal approaches are recommended by the CNGOF (grade C).

A new Medical Device (MD), the vNOTES (Vaginal Natural Orifice Transluminal Endoscopy System) offers the advantage of two approaches for pelvic surgery by allowing minimally invasive surgery to be performed by endoscopy through the vagina, offering perfect vision for the assistants and the operator and without scarring. Two randomized trials have shown that vNOTES allows, compared to laparoscopy, to perform adnexectomies and hysterectomies without conversion with less pain, fewer postoperative complications and a shorter hospitalization time.

The first evaluations of vNOTES are encouraging and suggest a new era for pelvic surgery: less postoperative pain, fewer complications and facilitation of ambulatory care. Also the videoscopic assistance of the vNOTES is a pedagogical tool for the vaginal route because the field of vision is no longer limited to the operator alone. However, the vNOTES has only been evaluated by the developers of the tool, in monocentric studies and in small numbers. The hysterectomy study evaluated only 35 patients with vNOTES, half of whom had a uterus of less than 280 g. The benefit of vNOTES for uteri smaller than 280 g is not obvious because of the ease of the surgical procedure and the cost of the "classic" vaginal route. Our study would be the first multicentric and academic study on vNOTES to focus specifically on large volume uteri, the most difficult to operate and prone to postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Any woman received in preoperative consultation in the Gynecology-Obstetrics Department for a benign pathology of a uterus estimated to be large requiring a hysterectomy.
* Patient affiliated or entitled to a social security system
* Patients over 18 years of age
* Patients having given their agreement to participate and after signing the consent form

Exclusion Criteria:

* Woman refusing to participate in the study (lack of consent)
* Non-French speaking woman (unable to conduct a good quality interview of the pregnant woman)
* Participation in another interventional study.
* Patient subject to a legal protection measure or unable to express her consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patient with complications | From surgery to 6 weeks of surgery
  The proportion of patients with at least one pre- and post-operative complication at 6 weeks will be estimated along with its 95% confidence interval in each surgical strategy group.
  The primary endpoint is a composite endpoint including the occurrence of intraoperative and postoperative complications within 6 weeks of surgery.
  Postoperative complications were Infectious complications, Bleeding complications and All hospital readmissions related to the procedure Postoperative complications will be classified according to the Clavien-Dindo classification
  Intraoperative complications will be defined as :
  * wounds of nearby organs (bladder, ureters, rectum, colon, small intestine)
  * and bleeding defined as bleeding requiring immediate resumption, intraoperative transfusion and/or decreasing the patient's hemoglobin by more than 2 points compared to the last known preoperative blood sample

SECONDARY OUTCOMES:
Conversion | During surgery
  Number of patients with conversion during surgery

OTHER OUTCOMES:
Post-operative pain | From surgery to 3 hours of surgery
  Maximal Pain measured by a numerical scale : 0 no pain / 10 maximum pain
Short-term postoperative pain | From surgery to 1 week after surgery
  Maximal short-term postoperative pain the first week after surgery measured by a numerical scale (0 no pain / 10 maximum pain) by a daily telephone call
Duration of postoperative reflex ileus | Day 0
  Duration of post-operative reflex ileus between the day of the operation and the resumption of a transit (appearance of the first gas) in hours
Duration of the operation | Surgery
  operative time will be evaluated between the incision and the end of the closure, in minutes.
Duration of hospitalization and the possibility of returning home | last day of hospitalization
  The length of hospital stay will be assessed in days and the possibility of return home by the time in hours from surgical incision to a Chung≥ score of 9/10. The Chung score assesses the possibility of a return home in ambulatory surgery.
Sexual dysfunction | 3 months
  Sexual disorders: sexual life will be assessed by the difference in the specific validated score (self-questionnaire) (PISQ12 with a score ranging from 0 to 48) between the inclusion date and 3 months after surgery for sexually active women.

CONTACTS AND LOCATIONS:
Overall Officials: Céline CHAULEUR, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (6):
- France (6):
  - HFME - Hospices Civils de Lyon, Bron
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Ch Issoire, Issoire
  - CHU LIMOGES - Hôpital de la mère et de l'Enfant, Limoges
  - CHU Saint-Etienne, Saint-Etienne
  - Clinique Mutualiste de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No